CLINICAL TRIAL: NCT02732041
Title: Asynchrony During Mechanical Ventilation in Patients With Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Responsible Party: Principal Investigator, Pablo Oscar Rodriguez, Assosiated Professor, Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Other Study IDs: CEMIC1008
Record Dates: First submitted 2016-03-19; First posted 2016-04-08 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Respiratory Distress Syndrome, Adult; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Asynchrony during mechanical ventilation has been poorly described in patients suffering from acute respiratory distress syndrome. The purpose of this study is to describe the frequency of asynchronies (ineffective efforts and double triggering) in these group and evaluate potential risk factors and prognosis implications.

DETAILED DESCRIPTION:
Major patient-ventilator asynchronies have been described during assisted mechanical ventilation in different settings. Few studies have evaluated double cycling in ARDS patient. No clear predictors of this finding beside low tidal volume have been found, and clinical outcome implications have not been addressed. This study has 3 main objectives: evaluate the frequency of double cycling and ineffective efforts, seek for potential predictors and clinical outcomes related to asynchronies. Subjects with less than 72 hours of mechanical ventilation due to ARDS will be recruited. Thirty minutes of mechanical ventilation will be recorded and automatically analyzed with a custom-made program to detect asynchronies. A blood sample will be drawn to measure inflammatory and lung tissue damage biomarkers. Clinical and outcome data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Acute Respiratory Distress Syndrome according to Berlin definition
* Intubation and mechanical ventilation within 72 hours of inclusion

Exclusion Criteria:

* Known severe neuromuscular disease
* Continuous neuromuscular blocking agents infusion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of acute respiratory distress syndrome and mechanical ventilation for less than 72 hours
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Asynchrony rate | 30 minutes
  Asynchronies per minutes of mechanical ventilation

SECONDARY OUTCOMES:
Length of mechanical ventilation | From the date of intubation to the date of complete weaning from mechanical ventilation or death which ever comes first, up to 90 days
ICU mortality | From the date of admission to the date of discharge from the ICU, up to 90 days
Hospital mortality | From the date of admission to the date of discharge from the ICU, up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Pablo O Rodriguez, MD, Principal Investigator — Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Locations (5):
- Argentina (5):
  - Complejo Medico Churruca Visca, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Sanatorio Anchorena, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Sanatorio La Trinidad Mitre, Ciudad Autonoma Buenos Aires, Buenos Aires
  - CEMIC (Centro de Educación Médica e Investigaciones Clínicas), CABA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez PO, Tiribelli N, Fredes S, Gogniat E, Plotnikow G, Fernandez Ceballos I, Pratto R, Raimondi A, Guaymas M, Ilutovich S, San Roman E, Madorno M, Maskin P, Brochard L, Setten M; Grupo Argentino de Estudio de Asincronias en la Ventilacion Mecanica Study Group. Prevalence of Reverse Triggering in Early ARDS: Results From a Multicenter Observational Study. Chest. 2021 Jan;159(1):186-195. doi: 10.1016/j.chest.2020.08.018. Epub 2020 Aug 14. PMID 32805238